CLINICAL TRIAL: NCT04729426
Title: The Effect of Using a Birthing Ball During Labor on the Labor Process
Brief Title: Birthing Ball (Peanut Ball) Positions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gonca Karataş Baran (Other)
Responsible Party: Sponsor-Investigator, Gonca Karataş Baran, Ankara Yildirim Beyazıt University Student, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AnkaraYBU sbe
Record Dates: First submitted 2021-01-23; First posted 2021-01-28 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Labor Pain; Labor Long
Keywords: Peanut ball; Birthing ball; labor positions; labor process
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: There will be two group. One is interventional group; other is control group.
Who Masked: Participant
Masking Description: The volunteer who is in the latent phase of labor will not know which group she will be in before joining the study. After accepting to participate in the study, the volunteer will be informed about which group she will be in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Position Group (Experimental): Position group
  Interventions: Other: Peanut Ball Position
- Control group (No Intervention): No Position group

INTERVENTIONS:
Other: Peanut Ball Position — The group of healthy pregnant women who meet the inclusion criteria will be determined by randomization according to the order of application to the delivery room. A group (intervention group) will be given positions using the peanut ball tool in active phase and transition phase and the positions will be changed every 30 minutes.
  Arms: Position Group

SUMMARY:
In this study, it was aimed to position by using peanut ball, which is a kind of birth ball, in the first stage of delivery in pregnant women who are planned to have vaginal delivery with cephalic admission, who is a primipara, who do not have a risky pregnancy and systemic disease; It will be done to determine the effect on the birth process.

DETAILED DESCRIPTION:
The group of healthy pregnant women who meet the inclusion criteria will be determined by randomization according to the order of application to the delivery room in the latent phase. Positions will be changed every 30 minutes using the peanut ball tool in a group (intervention group) in active phase and transition phase. These positions are; side-lying position, compressed side-lying position, semi-sitting position, forward leaning position, upright sitting position and pushing position. All positions will be given to the pregnant woman by the researcher and she will be with the pregnant woman during the position intervention. How to give the peanut ball positions is indicated in the flow chart with photographs. Position application will not be applied to the other group (control group), routine procedure of the hospital will be applied.

Parameters to Look for:

The researcher will evaluate the progress of the birth process (cervical dilatation and effacement, fetal head descent, Fetal Hearth Rate, duration of the first and second stages of labor), delivery method and information about the baby (gender, weight, height and head circumference length, APGAR) in both groups of women from the hospital's partograph records. Information on the progress of the birth process from the active phase of each pregnant birth to the completion of the birth process in the hospital is processed in the partograph with 30 minutes intervals.

The pain level in each stage and phases of labor will be evaluated by the researcher with a visual pain scale.

The first breastfeeding process will be observed and evaluated by the researcher using the "LATCH Breastfeeding Diagnostic and Evaluation Scale" in the delivery room.

Finally, when the mother relaxes physically and goes to bed, the researcher will apply the "Birth Satisfaction Scale" to assess maternal satisfaction with care at birth.

Study Group Population: The population of the study will be composed of primiparous pregnant women who applied to Ankara City Hospital Obstetrics and Gynecology Clinic Delivery Room.

Sample of the Study Group: Since there is no reference study (duration of delivery) for the main research question created to examine the difference in the intervention and control groups, the required sample size calculation will be made in groups of twenty (case: 20, control: 20) and the effect width will be calculated and Type I error 0.05 and it will be made with 95% power.

Since the minimum number of samples required is taken into account with loss, 20% will be added. The G power program will be used to calculate the number of samples required for the study.

The randomization of the groups for pre-application was done with the computer randomization program Random Allocation Software. Pre-application data will be included in the research data. The number of pregnant women in the pre-application will be subtracted from the number of pregnant women required according to the number of samples determined after the pre-application, and re-randomization for the remaining number of pregnant women will be made with this program.

Data Evaluation: The compatibility of the continuous variables to be obtained within the scope of the study to normal distribution will be examined with the Shapiro-Wilk test. Mean ± standard deviation will be used in the representation of descriptive statistics related to the variables that conform to the normal distribution, while the median (Interquartile Width - DIAG; minimum; maximum) will be used for distorted data, and the number and percentage will be used in the representation of categorical variables. In comparison of the variables measured in the groups, the necessary assumptions will be examined and appropriate t-test or Man-Whitney u test methods will be used. Comparison of groups and categorical variables will be made with the appropriate chi-square tests. All hypotheses will be established bilaterally and the statistical significance level will be accepted as p <0.05. IBM SPSS Statistics 23.0 program will be used for statistical analysis and calculations.

Data Collection Tools:

Data will be collected with the data collection form (Case Report Form). The data collection form consists of five parts.1. General Information;2. Observations and Findings;3. Visual Pain Scale;4. Birth Satisfaction Scale:5. LATCH Breastfeeding Diagnostic and Evaluation Scale.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous at 37-42 weeks of gestation,
* between the ages of 18-40,
* Not diagnosed with risky pregnancy (Intrauterine Growth Retardation, Fetal Anomaly, Polyhydramnios or Oligohydraamnios, Thromboembolic Diseases, Presentation Anomalies, Premature Membrane Rupture, Multiple Pregnancy, Sexually Transmitted Disease, Preeclampsia / Eclampsia etc.)
* Without systemic disease (Hypertension, Heart Disease, Diabetes, Asthma, Thyroid, Epilepsy, etc.)
* Single pregnancy,
* Vaginal delivery planned with cephalic admission,
* in the latent phase of labor,
* Epidural anesthesia / analgesia was not applied,
* Volunteering to participate in research,
* Pregnant women who do not have any communication disorder will be taken.

Exclusion Criteria:

* Failure to meet the inclusion criteria is the exclusion criteria.

Exclusion (Withdrawal) from the Study Criteria

* Having adaptation problems in applying the positions to be given,
* Maternal (vital signs deviation from normal, hyperstimulation, abnormal bleeding, etc.) and fetal complications (such as fetal distress, cord entanglement, cord prolapse) during delivery,
* Caesarean section, which could not complete the normal birth process,
* Pregnant women who give up working at any stage of the study will be excluded from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primipara pregnant woman
Enrollment: 101 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Labor time | max 8 hour
  Firsth stage ( active phase and transition phase) time+ and second stage labor time=...minutes

SECONDARY OUTCOMES:
cervical dilation | max 8 hour
  hourly cervical dilation findings
cervical effacement | max 8 hour
  hourly cervical effacement findings
fetal head level | max 8 hour
  hourly fetal head level findings
The pain level | max 8 hour
  The pain level in each stage and phases of labor will be evaluated by the researcher with visual pain scale.The pregnant woman marks her own pain on a 10 cm horizontal ruler with painlessness on one end of the scale and the most severe pain on the other . In the study conducted, the visual comparison scale of ten units will be evaluated as the level of pain experienced at birth: 0 = None, 10 = Intractable pain. Pain scale level categorization; It will be categorized in four sections as 0 points: no pain, 1-4 points: mild pain, 5-6 points: moderate pain, 7-10 points: severe pain.
The first breastfeeding process evaluation | within 30 minutes after labor
  The first breastfeeding process will be observed and evaluated by the researcher using the "LATCH Breastfeeding Diagnostic and Evaluation Scale" in the delivery room.The name of the diagnostic tool LATCH is derived from the English initials of these five criteria: L, Latch on the brest; A, seeing / hearing the baby's swallowing movement (Audible swallowing); T is the type of the nipple; C is the mother's comfort regarding the nipple and nipple (Comfort breast / nipple) and H is the holding position for the baby (Hold / Help). Each item is scored between 0-2 points. The total score that can be obtained from the tool is 0-10, and the high score means higher breastfeeding success.
maternal satisfaction | within 30 minutes to two hours after labor
  "Birth Satisfaction Scale" will be applied to evaluate maternal satisfaction with care at birth.Birth Satisfaction Scale is a measurement tool that consists of 10 items and has 3 sub-dimensions, applied to women who give normal birth in the first ten days postpartum.The scale is 5-point Likert type. Strongly disagree, "0 point", disagree "1 point", indecisive "2 points", agree "3 points", strongly agree "4 points". The scale is between 0 and 40 points. 6 items are positive, 4 items are negative, and 4 items are scored in reverse. The reverse scored items are 2., 4., 7, and 8. The higher the score obtained from the scale, the higher the birth satisfaction of the woman.

CONTACTS AND LOCATIONS:
Overall Officials: Esma SARIKAYA, professor, Study Director — Ankara City Hospital Bilkent
Locations (1):
- Ankara Şehir Hastanesi Kadın Doğum Hastanesi, Ankara, Bilkent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tussey CM, Botsios E, Gerkin RD, Kelly LA, Gamez J, Mensik J. Reducing Length of Labor and Cesarean Surgery Rate Using a Peanut Ball for Women Laboring With an Epidural. J Perinat Educ. 2015;24(1):16-24. doi: 10.1891/1058-1243.24.1.16. PMID 26937158
- [Result] Roth C, Dent SA, Parfitt SE, Hering SL, Bay RC. Randomized Controlled Trial of Use of the Peanut Ball During Labor. MCN Am J Matern Child Nurs. 2016 May-Jun;41(3):140-6. doi: 10.1097/NMC.0000000000000232. PMID 26859467
- [Result] Grenvik JM, Rosenthal E, Saccone G, Della Corte L, Quist-Nelson J, Gerkin RD, Gimovsky AC, Kwan M, Mercier R, Berghella V. Peanut ball for decreasing length of labor: A systematic review and meta-analysis of randomized controlled trials. Eur J Obstet Gynecol Reprod Biol. 2019 Nov;242:159-165. doi: 10.1016/j.ejogrb.2019.09.018. Epub 2019 Sep 20. PMID 31600716